CLINICAL TRIAL: NCT04384952
Title: Randomized Controlled Trial Comparing the Effect of a Parent-guided Speech and Language Therapy Program During the Summer Holidays With an Adapted Holiday Book on the Reading Level of Children With Visual-attentional Dyslexia
Brief Title: Effectiveness of a Parent-administered Reading Therapy Program During Summer Break for Dyslexic Children
Acronym: REEDVAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: APHP200214; IDRCB 2019-A03260-57 (Other: ANSM)
Record Dates: First submitted 2020-04-28; First posted 2020-05-12 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2020-04

CONDITIONS: Dyslexia
MeSH Terms: conditions — Dyslexia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parent-administered reading therapy. (Experimental): Parent-administered reading therapy program: 15min each day, 5 days a week during 6 weeks during the summer break. Repeated reading with feedback from the parent and time control.
  Interventions: Other: Parent-administered reading therapy.
- Dyslexic's Holliday Workbook. (Active Comparator): Use of a special Dys holiday book, no parent-guided training.
  Interventions: Other: Dyslexic's Holiday Workbook

INTERVENTIONS:
Other: Parent-administered reading therapy. — Parent-administered reading therapy program: 15min each day, 5 days a week during 6 weeks during the summer break. Repeted reading with feedback from the parent and time control.
  Arms: Parent-administered reading therapy.
Other: Dyslexic's Holiday Workbook — Use of a special Dyslexic's holiday book, no parent-guided training.
  Arms: Dyslexic's Holliday Workbook.

SUMMARY:
"After summer break, the reading performance of dyslexic children declines more than those of non-dyslexic children. Indeed, during the summer, dyslexic children are less inclined to read and their consultations with speech therapist are usually suspended.

Intensive speech therapy programs proved to be efficient during the summer, to maintain reading level of dyslexic children. However these programs are expensive and not easy to generalise. Some other studies tested reading therapy programs applied by parents at home. It proved to be effective and feasible.

Thus, the hypothesis of the present study is: a parent-administered reading therapy program during the summer break could stabilise the reading performance of dyslexic children after the summer. On the contrary the investigators assume the control group reading performance would decrease."

DETAILED DESCRIPTION:
"Dyslexia is a specific learning disability characterised by reading difficulties, not caused by developmental, neurological or sensory (vision or hearing) disorders.

After summer break, the reading performance of dyslexic children declines more than those of non-dyslexic children. Indeed, during the summer, dyslexic children are less inclined to read and their consultations with speech therapist are usually suspended.

Intensive reading therapy programs proved to be efficient during the summer, to maintain reading level of dyslexic children. However these programs are expensive and not easy to generalise. Some other studies tested reading therapy programs applied by parents at home. It proved to be effective and feasible.

Thus, the hypothesis of the present study is: a parent-administered reading therapy program during the summer break could stabilise the reading performance of dyslexic children (grade 3 to 5) after the summer. On the contrary the investigators assume the control group reading performance would decrease.

With a controlled randomised trial, the investigators will compare the reading performance of two groups of dyslexic children with the same type of dyslexia (with visual information treatment deficit). All of them are diagnosed by the Reference Centre for learning disabilities (CRTLA), a Robert Debré Hospital's Unit, Paris (France).

Intensity and duration : 6 weeks during the summer break. 15 minutes/day, 5 times per week.

Intervention group : Parent-administered reading therapy program. Control group : Dyslexic's Holiday Workbook (Hatier Editor). This study's main objective consists in evaluating the effectiveness in reading performance of a parent-administered reading training program during the summer break for dyslexic children.

"

ELIGIBILITY:
Inclusion Criteria:

* Schooled in Grade 3, 4 or 5 (CE2, CM1 ou CM2) at inclusion
* Diagnosis of developmental dyslexia with visual information treatment deficit, confirmed by the Reference Center for Learning Disabilities, Robert Debré Hospital
* Speech therapy for dyslexia that has started for at least 6 months
* No speech therapy during the 6-weeks intervention
* Family interest and availibility for 6 weeks durant summer break
* Informed consent signed by parents
* Affiliation to a social security scheme

Exclusion Criteria:

* Parents not fluent enough in French to read a text
* Patient IQ (intelligence quotient) < 70 (WISC test- Wechsler Intelligence Scale for Children)
* Other neurological pathology in the foreground
* Presenting hearing disorders or visual disorders not treated,
* Member of a sibling also eligible for the protocol (contamination bias)
* Beneficiary of State medical aid (AME)

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2020-06-05 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
Measuring program effectiveness on reading performance (accuracy and speed of word reading) | 4 weeks
  Word Reading performance with French BALE Test. BALE (Batterie Analytique du Langage Ecrit). Measure of number of correct words read and speed of reading. Raw score for word reading performance (accuracy) : minimum 0 (worse outcomme, maximum 20 (better outcome)

CONTACTS AND LOCATIONS:
Locations (1):
- Robert Debre Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Kerjean L, Benard P, Peyre H. Parent-implemented intervention for children in third to fifth grade with dyslexia. Encephale. 2023 Dec;49(6):589-595. doi: 10.1016/j.encep.2022.08.016. Epub 2022 Oct 15. PMID 36253171